CLINICAL TRIAL: NCT04215874
Title: Caudal Epidural Block and Ultrasound-guided Dorsal Penile Nerve Block With the In-plane Technique for Pediatric Distal Hypospadias Surgery: A Prospective Observational Study
Brief Title: Caudal Epidural Block and DPNB in Hypospadias
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Volkan Ozen, Principal Investigator, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: 2019/1219
Record Dates: First submitted 2019-12-28; First posted 2020-01-02 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Hypospadias; Postoperative Pain
Keywords: dorsal penile nerve block; caudal epidural block; postoperative pain; analgesia; hypospadias; ultrasound
MeSH Terms: conditions — Hypospadias; Pain, Postoperative; Agnosia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dorsal penile nerve block group: Ultrasound (US) guided dorsal penile nerve block with in plane technique was done.
  Half of the total 0.2 ml/kg dose of 0.25% bupivacaine was administered while observing its distribution with US. The same procedure was then repeated on the other side of the penis.
- Caudal epidural block group: A 22 G needle was inserted through the sacral hiatus. The loss of resistance method was used to pass through the sacrococcygeal membrane and enter the caudal epidural space. Negative aspiration was then performed 0.25% bupivacaine at a dose of 0.2 ml/kg was administered.

SUMMARY:
Hypospadias, seen in every 200-300 births, is one of the most common congenital anomalies of the penis and is defined as the urethral meatus being located in the ventral part of the penis instead of its normal place. The surgery of this anomaly is very painful in the postoperative period and requires long-term analgesia. Regional anesthesia methods combined with general anesthesia play an important role in providing effective and long-term postoperative pain control in pediatric penile surgery. These methods also reduce postoperative morbidity, enable early mobilization and significantly decrease the need for narcotic analgesics.

The investigator's hypothesis is peripheral nerve blocks are superior to neuraxial blocks as the blocks provide longer-term analgesia and have fewer side effects.

DETAILED DESCRIPTION:
The surgery of hypospadias is very painful in the postoperative period and requires long-term analgesia. A dorsal penile nerve block (DPNB) and caudal epidural block (CEB) are commonly used regional anesthesia techniques for postoperative pain control.

Aims: The primary aim of the current study was to use the duration until the first postoperative analgesic requirement after two different block techniques to compare the analgesic effect. The secondary aims were to compare the two methods for postoperative Children's Hospital Eastern Ontario Pain Scale (CHEOPS) scores, complications and parental satisfaction scores.

ELIGIBILITY:
Inclusion Criteria:

* 1-7 years of age
* ASA (American Society of Anesthesiologists) I-II group
* Scheduled for distal hypospadias surgery
* Able to communicate in Turkish
* Willing to participate to the study (parents and children)

Exclusion Criteria:

* Less than 1 or more than 7 years of age
* A neurological deficit, bleeding diathesis, or a history of local anesthetic allergy; an infection or redness in the injection area, congenital low back anomaly, liver disorder, a psychiatric disorder, mental retardation, or communication problems detected during examination
* Unwilling to to participate to the study ((parents or children)

Ages: 1 Year to 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: The study was conducted with children who underwent hypospadias surgery at a training and research hospital in Istanbul, Turkey.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2019-04-14 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Time of Postoperative analgesic requirement | Up to 24 hours
  It was assessed six times after the operation with Children's Hospital Eastern Ontario Pain Scale. The lowest scale score is 4 points and the highest 13 points. Significant pain behavior for Children's Hospital Eastern Ontario Pain Scale has been identified as 7 points or more. Following transfer from the recovery unit to the ward, the 1st, 2nd, 6th, 12th and 24th hour pain levels were evaluated by the ward nurse. Paracetamol was administered IV at a dose of 10 mg/kg if the scale score was 7 or higher.

SECONDARY OUTCOMES:
Level of Postoperative pain | Up to 24 hours
  It was assessed six times after the operation with Children's Hospital Eastern Ontario Pain Scale. The lowest scale score is 4 points and the highest 13 points. Significant pain behavior for Children's Hospital Eastern Ontario Pain Scale has been identified as 7 points or more. Following transfer from the recovery unit to the ward, the 1st, 2nd, 6th, 12th and 24th hour pain levels were evaluated by the ward nurse.
Rate of Postoperative complications | Up to 24 hours
  Urinary retention, nausea, vomiting, lower extremity numbness, motor block were postoperative complications. They were assessed by ward nurse.
Level of Parent satisfaction | Up to 24 hours
  The parents were asked about their satisfaction with the child's comfort and activity level [1, unsatisfied; 2, satisfied (good); 3, absolutely satisfied (excellent)] at the 24-hour follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Volkan Ozen, MD, Study Director — Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Locations (1):
- Okmeydani Training and Research Hospital, Istanbul, Şişli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alizadeh F, Heydari SM, Nejadgashti R. Effectiveness of caudal epidural block on interaoperative blood loss during hypospadias repair: A randomized clinical trial. J Pediatr Urol. 2018 Oct;14(5):420.e1-420.e5. doi: 10.1016/j.jpurol.2018.03.025. Epub 2018 May 21. PMID 29858133
- [Background] Kundra P, Yuvaraj K, Agrawal K, Krishnappa S, Kumar LT. Surgical outcome in children undergoing hypospadias repair under caudal epidural vs penile block. Paediatr Anaesth. 2012 Jul;22(7):707-12. doi: 10.1111/j.1460-9592.2011.03702.x. Epub 2011 Sep 29. PMID 21957982
- [Background] Suleman MI, Akbar Ali AN, Kanarek V, Li M, Patel A. Ultrasound Guided In-Plane Penile Nerve Block for Circumcision: A New, Modified Technique Suggests Lower Anesthetic Volume and Narcotic Use. Middle East J Anaesthesiol. 2016 Oct;23(6):647-53. PMID 29939703
- [Derived] Ozen V, Yigit D. Caudal epidural block versus ultrasound-guided dorsal penile nerve block for pediatric distal hypospadias surgery: A prospective, observational study. J Pediatr Urol. 2020 Aug;16(4):438.e1-438.e8. doi: 10.1016/j.jpurol.2020.05.009. Epub 2020 May 20. PMID 32507565